CLINICAL TRIAL: NCT00006463
Title: Phase I Study of ET-743 in Pediatric Refractory Solid Tumors
Brief Title: Ecteinascidin 743 in Treating Children With Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P9972; COG-P9972 (Other: Children's Oncology Group); POG-P9972 (Other: Pediatric Oncology Group); CDR0000068273 (Other: Clinical Trials.gov)
Record Dates: First submitted 2000-11-06; First posted 2004-04-26 (Estimated); Last update posted 2014-02-21 (Estimated); Status verified 2014-02

CONDITIONS: Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: unspecified childhood solid tumor, protocol specific
MeSH Terms: interventions — Trabectedin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Therapy ECTEINASCIDIN 743 (1100 ug/m2 ) (Experimental)
  Interventions: Drug: ECTEINASCIDIN 743
- ECTEINASCIDIN 743 (1300 ug/m2) (Experimental)
  Interventions: Drug: ECTEINASCIDIN 743

INTERVENTIONS:
Drug: ECTEINASCIDIN 743
  Other Names: ET-743; NSC S648766; IND 50,286

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Ecteinascidin 743 may be an effective treatment for solid tumors.

PURPOSE: Phase I trial to study the effectiveness of ecteinascidin 743 in treating children who have refractory solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose and dose-limiting toxicity of ecteinascidin 743 in pediatric patients with refractory solid tumors. II. Determine the pharmacokinetics of this drug in these patients. III. Determine the antitumor activity of this drug in this patient population.

OUTLINE: This is a dose escalation, multicenter study. Patients are stratified according to pretreatment (pretreated vs less heavily pretreated). Patients receive ecteinascidin 743 IV over 3 hours on day 1. Treatment continues every 3 weeks in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of ecteinascidin 743 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicities.

PROJECTED ACCRUAL: A total of 3-20 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed malignant solid tumor at original diagnosis Refractory to standard treatment or no curative therapy available No CNS tumor No bone marrow metastases (for less heavily pretreated stratum only)

PATIENT CHARACTERISTICS: Age: At least 365 days to 17 years Performance status: Karnofsky 50-100% (for patients older than 10 years) Lansky 50-100% (for patients 10 years and younger) Life expectancy: At least 8 weeks Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 (transfusion independent) Hemoglobin at least 8.0 g/dL (RBC transfusion allowed) Hepatic: Bilirubin no greater than normal SGPT no greater than 2.5 times normal Albumin at least 2 g/dL Alkaline phosphatase normal Gamma glutamyl transferase less than 2.5 times normal Renal: Creatinine no greater than 1.5 times normal OR Creatinine clearance or GFR at least lower limit of normal Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception Creatine phosphokinase less than 2 times normal No uncontrolled infection Seizure disorder allowed if well controlled on anticonvulsants No CNS toxicity greater than grade II

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 1 week since prior biologic therapy and recovered At least 1 week since prior growth factor therapy At least 6 months since prior peripheral blood stem cell transplantation and no evidence of graft-vs-host disease For less heavily pretreated stratum: No prior peripheral blood stem cell transplantation Chemotherapy: At least 4 weeks since prior myelosuppressive chemotherapy (6 weeks for nitrosoureas) and recovered No prior ecteinascidin 743 For less heavily pretreated stratum: No more than 2 prior chemotherapy regimens Endocrine therapy: Not specified Radiotherapy: At least 2 weeks since prior local palliative radiotherapy (small port) At least 6 weeks since prior substantial bone marrow radiotherapy At least 6 months since prior craniospinal radiotherapy or radiotherapy to 50% or greater of pelvis For less heavily pretreated stratum: No prior craniospinal irradiation of 18Gy or greater No prior irradiation to greater than 50% of pelvis Recovered from toxic effects of prior radiotherapy Surgery: Not specified Other: No concurrent foods or medication that interferes with P-450 metabolism Anticonvulsants allowed

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2000-10; Primary Completion 2005-01 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | Length of study

SECONDARY OUTCOMES:
Dose Limiting Toxicity
  To determine the maximum tolerated dose (MTD) of vincristine, when used in combination with irinotecan, and the dose-limiting toxicity (DLT) of this combination; irinotecan will be administered IV over 1 hour x 5 days, q 21 days, with vincristine IVP days 1, 8, 15, 22, 29, every 42 days, to children with refractory solid tumors.
Determine a safe and tolerable dose of vincristine, when administered with irinotecan
  To determine a safe and tolerable dose of vincristine, when administered with irinotecan, for future evaluation in phase II clinical trials.
Determine the pharmacokinetics of vincristine and irinotecan | Length of study
  To determine the pharmacokinetics of vincristine and irinotecan (and its active metabolite SN-38) when administered in combination to children with refractory cancer.
Determine the incidence and severity of other toxicities | Length of study
  To determine the incidence and severity of other toxicities of this combination.
Seek preliminary evidence of anti-tumor activity of irinotecan plus vincristine | Length of study
  To seek preliminary evidence of anti-tumor activity of irinotecan plus vincristine against recurrent solid tumors.

CONTACTS AND LOCATIONS:
Overall Officials: Sylvain Baruchel, MD, Study Chair — The Hospital for Sick Children
Locations (47):
- United States (42):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - University of California San Diego Cancer Center, La Jolla, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Beckman Research Institute, City of Hope, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital at Stanford, Palo Alto, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Shands Hospital and Clinics, University of Florida, Gainesville, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - Children's Memorial Hospital, Chicago, Chicago, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - Boston Floating Hospital Infants and Children, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospital, Kansas City, Missouri
  - Cardinal Glennon Children's Hospital, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Columbia Presbyterian Hospital, New York, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Children's Hospital Medical Center - Cincinnati, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt Cancer Center, Nashville, Tennessee
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Australia (2):
  - Royal Children's Hospital, Parkville, Victoria
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (3):
  - Hospital for Sick Children, Toronto, Ontario
  - Montreal Children's Hospital, Montreal, Quebec
  - Hopital Sainte Justine, Montreal, Quebec

REFERENCES:
- [Result] Lau L, Supko JG, Blaney S, Hershon L, Seibel N, Krailo M, Qu W, Malkin D, Jimeno J, Bernstein M, Baruchel S. A phase I and pharmacokinetic study of ecteinascidin-743 (Yondelis) in children with refractory solid tumors. A Children's Oncology Group study. Clin Cancer Res. 2005 Jan 15;11(2 Pt 1):672-7. PMID 15701855